CLINICAL TRIAL: NCT03326765
Title: Characterizing Sleep Disorders in Children and Adults With Tuberous Sclerosis Complex (TSC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Study coordinator, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: TSC v 1.0
Record Dates: First submitted 2017-10-06; First posted 2017-10-31 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Sleep Disorder
Keywords: tuberous sclerosis complex (TSC); Children; Adults
MeSH Terms: conditions — Sleep Wake Disorders; Tuberous Sclerosis | interventions — Surveys and Questionnaires; Actigraphy

STUDY DESIGN:
Intervention Model Description: 2 groups:
  * 30 Children(0-18y) withTSC without epilepsy
  * 30 Adults(>18y) withTSC without epilepsy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children (Other): Questionnaires electroencephalogram (EEG) Actigraphy polysomnography
  Interventions: Other: Questionnaires; Procedure: electroencephalogram (EEG); Procedure: polysomnography; Procedure: Actigraphy
- Adults (Other): Questionnaires electroencephalogram (EEG) Actigraphy polysomnography
  Interventions: Other: Questionnaires; Procedure: electroencephalogram (EEG); Procedure: polysomnography; Procedure: Actigraphy

INTERVENTIONS:
Other: Questionnaires — * Epworth sleepiness scale
  * Pittsburgh sleep quality Index (PSQI)
  * EQ-5D Adults
  * Pediatric Daytime Sleepiness scale (PDSS)
  * Sleep disturbance Scale for Children (SDSC
  * EQ-5D Children
  * Sleaping diary
Procedure: electroencephalogram (EEG) — is an electrophysiological monitoring method to record electrical activity of the brain
Procedure: polysomnography — type of sleep study, is a multi-parametric test used in the study of sleep and as a diagnostic tool in sleep medicine
Procedure: Actigraphy — type of sleep study based on bracelet around the wrist

SUMMARY:
The proposed research project is aimed at further characterization of sleep problems and evaluation of their impact in children and adults with TSC, excluding epilepsy as contributing factor. Questionnaire-based studies have shown that sleep problems occur in up to half of the children and a third of adults with tuberous sclerosis complex (TSC). However, there is only limited information on the nature of sleep problems and their impact on patients with TSC and their families.

DETAILED DESCRIPTION:
Questionnaire-based studies have shown that sleep problems occur in up to half of the children and a third of adults with tuberous sclerosis complex (TSC). However, there is only limited information on the nature of sleep problems and their impact on patients with TSC and their families. It is known from a questionnaire-based study in children with TSC that they often wake early or wake frequently during the night, and that they can be more tired during the day. In some children, sleep-problems seem to be related to the presence of seizures during the night. This has been confirmed in a study on 10 children with TSC and epilepsy by a combination of polysomnography (sleep study) and electroencephalography (EEG). A questionnaire-based study in adults also revealed the association with epilepsy features, and showed influence of mental health complaints on sleep.

Sleep structure and quality will be assessed through formal sleep studies (polysomnography and actigraphy). The influence of abnormal brain activity on sleep will be mapped by simultaneous recording of brain activity by means of EEG. The impact of sleep disorders will be determined through interviews with individuals with TSC and their relatives. The investigators will also use questionnaires and diaries to supplement their findings.

Importance: It is expected that the results of this study will 1) improve our understanding of sleep problems in TSC, 2) provide additional information on the influence of TSC on sleep, 3) give a more in-depth view on the impact of sleep problems on the lives of individuals with TSC and their families, 4) increase awareness about sleep problems in TSC, and 5) contribute to a better management of sleep problems by patients and families.

ELIGIBILITY:
Inclusion Criteria:

Children and adults with definite TSC based on the 2012 Consensus Conference Diagnostic

Exclusion Criteria:

* daily alcohol intake
* pregnancy
* caffeine abuse (>4 cups/day)
* shift work
* drug abuse
* anti-depressive therapy
* medications as benzodiazepine, melatonin, phenobarbital and antihistamines
* the presence of clinical or electrographic seizures.

Ages: 1 Day to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-09-27 (Actual); Primary Completion 2019-11-01 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
characterize the sleep phenotype of TSC in children and adults without epilepsy | 1 night
  - Sleep efficiency (SE%): the percentage ratio between total sleep time and time in bed (TST/TIB*100)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Jansen, PhD, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Sonia De Weerdt, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Alessandra Pereira,, PhD, MD, Principal Investigator — Department of Pediatrics School of Medicine, PUCRS, Brazil; Magda Nunes, PhD, MD, Principal Investigator — Director, School of Medicine, PUCRS, Brazil; Brain Instititute of Rio Grande do Sul, Brazil; Oliviero Bruni, PhD, MD, Principal Investigator — Department of Developmental and Social Psychology, Sapienza University of Rome, Italy; Paolo Curatolo, PhD, MD, Principal Investigator — Director, Child Neurology and Psychiatry Unit, Systems Medicine Department, Tor Vergata University of Rome, Italy
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium